CLINICAL TRIAL: NCT03275584
Title: Sûreté de la Perfusion Myocardique Par la Tomographie d'émission Par Positron Avec l'Ammoniaque marqué au N-13 du Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Brief Title: Safety of PET MPI Using the CRCHUM N-13 Ammonia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17.015
Record Dates: First submitted 2017-09-04; First posted 2017-09-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: N-13 Ammonia Safety
Keywords: positron emission tomography; NH3

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Main arm (Experimental): N-13 ammonia intravenous injection; 2 injections, 3-7 MBq/kg per injection
  Interventions: Drug: N-13 ammonia intravenous injection

INTERVENTIONS:
Drug: N-13 ammonia intravenous injection — Participants will receive two injections of N-13 ammonia, once at "rest" and once at "stress" before undergoing positron emission tomography myocardial perfusion imaging

SUMMARY:
Positron emission tomography (PET) myocardial perfusion imaging (MPI) is an examination that helps to assess the function and perfusion of the heart. Completion of this examination requires the injection of a small dose of a radiotracer (a radioactive substance).

PET MPI is a state-of-the-art non-invasive cardiac imaging tool. The main goal of the PET MPI examination is to assess if one or more of the arteries feeding blood to your heart are blocked. This examination replaces an older technology (single photon emission computed tomography, or SPECT), and allows the obtention of more accurate information, and new information that the older SPECT technology did not assess. The radiation dose received as part of the procedure is also smaller with PET versus SPECT.

One of the substances which can be used for PET MPI is called N-13 ammoniac (NH3). For this clinical study, NH3 which will be produced at the Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), per the standards and methods prescribed by Health Canada. NH3 is not currently approved for clinical use by Health Canada. It is thus considered and experimental substance in the context of this study.

Participants will undergo PET MPI with the CRCHUM NH3. The PET MPI procedure itself is not an experimental procedure and is not part of the research protocol. Only the use of NH3 produced at the CRCHUM is experimental.

The main objective of this research study is to validate the production process and assess the safety of the NH3 produced at the CRCHUM cyclotron. Secondary objectives include the assessment of prescription practices amongst physicians who refer patients for PET MPI, and how they will change over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient being referred for clinically indicated positron emission tomography myocardial perfusion imaging at the Centre hospitalier de l'Université de Montréal

Exclusion Criteria:

* Pregnant women
* Claustrophobic patient unable to undergo the examination
* Breastfeeding women unwilling to temporarily stop breastfeeding
* Patient with contra-indication to: dipyridamole, aminophylline, dobutamine or exercise stress test (depending on the method of cardiovascular stress test chosen)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Adverse reaction to the N-13 ammonia injection | 1 hour
  The absence or presence of adverse reactions related to the N-13 ammonia injection, as a simple yes or no.
  The following tools will be used to establish the presence/absence of adverse reaction:
  * Questionnaire during and after the procedure
  * Vital signs monitoring before, during and after the procedure
  * Patient's self-reported side-effects from the procedure

SECONDARY OUTCOMES:
Incidence of specific adverse reactions to N-13 ammonia injection | 1 hour
  If any adverse reactions to the N-13 ammonia injection are reported (see Primary Outcome), the incidence of specific adverse reactions will be recorded and calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Juneau, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'université de Montréal, Montreal, Quebec, Canada